CLINICAL TRIAL: NCT05593393
Title: A Long-term Follow-up Cohort Study in Patients With Intraductal Papillary Mucinous Neoplasm
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Hospital (Other Government); Tongji Hospital (Other); The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Wu Xi, associate professor, Peking Union Medical College Hospital
Other Study IDs: K2378
Record Dates: First submitted 2022-10-21; First posted 2022-10-25 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: IPMN, Pancreatic
Keywords: IPMN; clinical outcomes; EUS
MeSH Terms: conditions — Pancreatic Intraductal Neoplasms | interventions — Endosonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Baseline sample includes 20ml blood sample, 1 oral flora swab and 1 stool sample.
  Follow-up samples include 10mL blood sample and remaining samples of pancreatic puncture tissue and/or cyst fluid during EUS
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Endoscopic ultrasound — The EUS follow-up will be conducted at baseline and every 12 months thereafter. For patients with new WF or HRS in the evaluation, the follow-up physician and the patient can jointly decide whether to perform EUS evaluation in the 6 or 3 month intensive follow-up.

SUMMARY:
Study objective: To establish a long-term follow-up cohort of patients with IPMN, study the follow-up, clinical outcomes and prognostic factors of patients with IPMN, and provide a basis for clinical decisions and guidelines.

Study design: This is a real world, multicenter, prospective, observational cohort study

DETAILED DESCRIPTION:
Baseline assessment will be conducted on IPMN patients who meet the inclusion conditions and are included in the study with informed consent, including: ① demographic characteristics (such as age, gender, etc.); ② Clinical features (such as symptoms, complications, past history, family history, living/eating habits); ③ Characteristics of laboratory indicators (such as pancreatic function, liver enzyme, bile duct enzyme, CA199, CEA in blood; CA199, CEA in cystic fluid, etc.); ④ Imaging features * (such as multiple or single lesions, diameter of cyst, whether there are mural nodules, diameter of main pancreatic duct, etc.); ⑤ Endoscopic ultrasound (EUS) features * (such as: cyst location, echo, maximum diameter, whether the cyst wall is thickened, wall nodules, the connection between the cyst and the main pancreatic duct, laser confocal endoscopy features, etc.); ⑥ Pathological information (cytology of cystic fluid; cytological smear of cystic lesion puncture, histopathology); ⑥ Molecular characteristics of cyst fluid (such as proteomics/mass spectrometry, new biomarkers, next generation sequencing (NGS), flora characteristics, etc.); ⑦ Treatment information (such as current medication, whether to have received endoscopic treatment, etc.).

The follow-up contents include: outpatient follow-up (symptoms, laboratory indicators; keeping peripheral blood samples) every six months;, imaging follow-up (including enhanced pancreatic MR and EUS imaging; the first pancreatic MRI follow-up was conducted 6 months after enrollment to determine the stability of the lesions) at baseline and every 12 months thereafter.

During the follow-up, if the patient died of various causes, the follow-up will be terminated; If enhanced nuclear magnetic resonance imaging or EUS imaging of the pancreas indicates worrisome features (WFs) or high-risk features (High risk stigmata, HRS), EUS-FNA ± nCLE should be performed (when performing EUS, perform contrast-enhanced ultrasonography on cystic lesions with mural nodules, and collect cystic fluid when puncturing some cystic lesions with sufficient volume).

If the cytological/histological pathological results of FNA indicate cancer or high grade dysplasia (HGD), or/and cystic fluid cytological results are positive, surgical treatment is recommended; If the FNA and cyst fluid cytology results are negative, the patients with WF will be followed up 6 months later, while the HRS patients will be followed up 3 months later (whether to accept EUS examination is decided jointly by the follow-up physician and the patient). It is suggested to review EUS-FNA ± nCLE according to the imaging results. If the patient was advised to receive surgical treatment due to IPMN, the follow-up was terminated.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years old or above;
2. Diagnosis: Imaging examination showed the presence of intraductal papillary mucinous cystic tumor (IPMN) without high-risk features (including WF and HRS);
3. The patient or family members can understand the study protocol, are willing to participate in the study, and provide written informed consent.

Exclusion Criteria:

1. The patient's clinical, imaging and auxiliary examination characteristics conform to the surgical indications of the International Association of Pancreatic Diseases (IAP) 2018 guidelines, and the patient has no surgical contraindication;
2. Previous history of pancreatic malignant tumor;
3. There were the following worrisome features (WF) of IPMN found in the past examination: acute pancreatitis, cyst size ≥ 30mm, cyst wall thickening/strengthening, main pancreatic duct diameter of 5-9.9mm, non enhanced mural nodules, sudden change of main pancreatic duct diameter with distal pancreatic atrophy;
4. The following high risk features of IPMN (HRS) were found in the past: obstructive jaundice, enhanced mural nodules or related solid components, and main pancreatic duct>10mm;
5. The patient or family member could not understand the conditions and objectives of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IPMN patients in Peking Union Medical College Hospital and other related research centers
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The termination of the follow-up of IPMN patients, including death termination and recommended surgery termination. | 3 years
  Patient died or was recommended for surgical treatment.

SECONDARY OUTCOMES:
The new development of worrisome features or high-risk stigmata | 3 years
  High-risk stigmata refers to obstructive jaundice, enhancing mural nodules or an associated solid component, and those with an MPD ≥10 mm. Worrisome features refer to acute pancreatitis, cyst size ≥30 mm, thickened/enhancing cyst wall, MPD measuring 5-9.9 mm, nonenhancing mural nodules, and abrupt change in MPD caliber with distal atrophy of the pancreatic gland.

CONTACTS AND LOCATIONS:
Overall Officials: Xi Wu, M.D., Study Director — Peking Union Medical College Hospital; Shengyu Zhang, M.D., Principal Investigator — Peking Union Medical College Hospital; Yiran Su, MD candidate, Principal Investigator — Peking Union Medical College Hospital